CLINICAL TRIAL: NCT04265404
Title: Prospective Evaluation of qSOFA (Quick Sequential Organ Failure Assessment Score) to Detect Systemic Infection in Neurosurgical Patients
Brief Title: Evaluation of qSOFA in Neurosurgical Patients
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Elisabeth H. Adam, Principal Investigator, Goethe University
Other Study IDs: 75/18
Record Dates: First submitted 2019-10-16; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Brain Injuries; Brain Trauma; Subarachnoid Hemorrhage
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to look if Quick Sequential Organ Failure Assessment Score score in detecting a eary Sepsis is afflicted by neurosurgical disorders

ELIGIBILITY:
Inclusion Criteria: one of the following diseases

* Subarachnoidal Bleeding
* Traumatic brain injury
* Spondylodiszitis

Exclusion Criteria:

* intubated before income
* Age under 16

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients brought to the ICU with Inclusion Citeria.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Baseline measurement of qSOFA at admission to ICU | Measurement at the time of admission to the intensive care unit
  assessment of qSOFA (Quick Sequential Organ Failure Assessment Score)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Konczalla, Prof., Principal Investigator — Johann Wolfgang Goethe Universität
Locations (1):
- Johann Wolfgang Goethe Universität, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided